CLINICAL TRIAL: NCT07114484
Title: The Accuracy of Artificial Intelligence in the Detection of Bifid Mandibular Canal on CBCT: A Diagnostic Accuracy Study
Brief Title: Accuracy of AI in Detecting Bifid Mandibular Canal on CBCT: A Diagnostic Accuracy Study
Acronym: BMC-AI
Status: Completed | Type: Observational
Sponsor: Sara Reda Abdelhamid Aboseif (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Sara Reda Abdelhamid Aboseif, Resident, Department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo University
Organization: Cairo University (Other)
Other Study IDs: OMFR-8-1-1
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: Bifid Mandibular Canal
Keywords: Bifid Mandibular Canal; Cone-Beam Computed Tomography; Artificial Intelligence; Deep Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT Images of mandibular canal: Diagnostic Test: Deep Learning-Based Model A deep learning-based diagnostic tool developed by a computer science expert. The model is built upon a convolutional neural network architecture and trained using our study datasets.
  Alternative Names:
  Artificial Intelligence (AI) Tool

SUMMARY:
The goal of this observational study is to evaluate how accurately a deep learning-based artificial intelligence (AI) model can detect and segment bifid mandibular canals (BMCs) on cone-beam computed tomography (CBCT) scans in Egyptian patients. This condition is a key anatomical variation that, if missed, may cause surgical complications such as nerve injury.

The study uses previously collected CBCT scans of individuals aged 15 and older from the Oral and Maxillofacial Radiology Department at Cairo University. The scans will be analyzed retrospectively.

The main questions it aims to answer are:

How closely does the AI model's segmentation of the mandibular canal match the expert manual segmentation?

How accurate is the AI model in identifying the presence or absence of bifid mandibular canals?

Participants are not actively involved. Instead, anonymized CBCT data will be analyzed using the AI model and compared to expert annotations to measure diagnostic performance.

DETAILED DESCRIPTION:
This retrospective diagnostic accuracy study aims to evaluate the performance of a novel artificial intelligence (AI) model in the segmentation and detection of bifid mandibular canals (BMC) on cone-beam computed tomography (CBCT) scans. The study will be conducted on anonymized DICOM data collected from a dental radiology archive, with no direct patient contact or intervention.

Study Rationale and Background Accurate identification of bifid mandibular canals is crucial for avoiding complications during oral surgical procedures. Manual identification on CBCT by experts is the current standard, yet it is time-consuming and subject to interobserver variability. Deep learning-based models have the potential to offer automated, reproducible, and efficient alternatives.

AI Model and Methodology The AI model used in this study will be developed using a 3D U-Net architecture implemented in the MONAI framework. Manual segmentation of mandibular canals, including bifid variants, will be performed using 3D Slicer software to serve as ground truth data. The AI model will be trained and validated using this ground truth.

Technical Workflow Data Collection: Retrospective DICOM CBCT images will be extracted and anonymized.

Manual Segmentation: Gold standard segmentation will be performed manually by an expert using 3D Slicer.

Model Development: The 3D U-Net model will be developed and trained using the MONAI framework in Python.

Evaluation: The trained model will be evaluated on unseen test data and compared to manual segmentation using standard performance metrics (Dice Similarity Coefficient, sensitivity, specificity, and accuracy).

Statistical Analysis: The Dice score will be used as the primary metric of agreement. Sample size was calculated based on expected performance values. Confidence intervals were computed, and statistical significance was assessed.

Sample Size Assessment A power calculation was conducted based on the sensitivity and specificity of the model using normal approximation methods. The total sample size was determined to ensure reliable performance evaluation with adequate power and precision.

Data Quality Assurance and Handling A structured process will be employed to ensure that CBCT scans used are of sufficient diagnostic quality.

All manual segmentations will be reviewed by a second radiologist to reduce bias.

All model outputs will be verified against the manual ground truth by a blinded expert.

Data inconsistencies, if present, will be flagged, documented, and excluded from the analysis.

Missing Data Management Given the retrospective nature, no missing data will be filled in or replaced because only complete and usable scans will be included in the study.

Statistical Plan The primary analysis will involve evaluating the overlap between the AI model and expert segmentations using the Dice coefficient. Secondary measures will include the sensitivity and specificity of the AI model in detecting bifid branches. All statistical analyses will be performed using Python libraries such as SciPy and NumPy.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans for Egyptian people older than 15 years old (both male and female subjects are to be included)
* The field of view of the selected scans should clearly show at least one mandibular canal completely (from the mandibular foramen to the mental foramen)

Exclusion Criteria:

* CBCT images of sub-optimal quality or artifacts/high scatter interfering with the proper assessment of the mandibular canal course.
* CBCT scans showing significant mandibular deformities.
* CBCT scans showing severe bone loss that extends to the mandibular canal.

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: CBCT scans were retrospectively collected from the database of the Oral and Maxillofacial Radiology Department at Cairo University. The population included adult patients who had previously undergone CBCT imaging for diagnostic purposes unrelated to bifid mandibular canal suspicion. The cases were selected to include both males and females from a diverse patient base representative of the general outpatient population attending the university dental hospital.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Segmentation accuracy of deep learning model compared to manual ground truth | immediately after the intervention
  Evaluation of the similarity between the AI-generated segmentation of the mandibular canal and the expert manual segmentation using the Dice similarity coefficient.

SECONDARY OUTCOMES:
Diagnostic accuracy of the AI model in detecting bifid mandibular canals | immediately after the intervention
  Assessment of the AI model's ability to correctly classify the presence or absence of bifid mandibular canals on CBCT scans compared to expert radiologists' detection. Binary output will be measured as Present or Absent, and performance will be evaluated using sensitivity, specificity, PPV, NPV, and accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Anter, Ph.D, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data, including raw CBCT scans and manual segmentations, will not be shared to protect patient confidentiality and comply with institutional ethics policies. Aggregated performance metrics are available upon reasonable request.